CLINICAL TRIAL: NCT01352078
Title: The Wound Etiology and Healing Study
Brief Title: Wound Etiology and Healing Study
Acronym: WE-HEAL
Status: Completed | Type: Observational
Sponsor: George Washington University (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Victoria Shanmugam, MD, Professor, George Washington University
Other Study IDs: 041408; KL2RR031974 (NIH); UL1RR031975 (NIH); R01NR013888 (NIH)
Record Dates: First submitted 2011-05-10; First posted 2011-05-11 (Estimated); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Wounds; Hidradenitis Suppurativa; Hidradenitis; Acne Inversa
Keywords: Non healing ulcer; Wound; Hidradenitis suppurativa; Acne Inversa; Hidradenitis
MeSH Terms: conditions — Wounds and Injuries; Hidradenitis Suppurativa; Hidradenitis

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. Residual tissue left over after routine debridement surgery
  2. Wound fluid that would otherwise be discarded
  3. Residual blood/ serum samples left over after pre-surgery blood tests have been performed.
  4. Wound biofilm
  5. Wound photographs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non Healing Ulcer
- Hidradenitis suppurativa

SUMMARY:
The purpose of the WE-HEAL Study is to help researchers use human tissue samples and health records to study the reasons why some patients heal quickly and some have problems healing wounds. All patients seen with an open wound or hidradenitis suppurativa are invited to participate. Information from this research may help to understand how to prevent and treat certain diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18
2. Open wound or hidradenitis suppurativa
3. English speaking
4. Able to give informed consent

Exclusion Criteria:

1. Non-English speaking.
2. Unable to give informed consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non healing wounds or hidradenitis suppurativa
Sampling Method: Non-Probability Sample
Enrollment: 743 (Actual)
Dates: Start 2011-05; Primary Completion 2022-01 (Actual); Study Completion 2022-01 (Actual)

PRIMARY OUTCOMES:
Time to wound healing | 10 years
  This prospective study will establish a biobank for collection of residual biopsy tissue discarded after debridement, and collection of other biospecimens at the discretion of the investigators including wound fluid and serum samples. Patients will also permit linking of biosamples to clinical outcomes data. Using a primary outcome of wound healing we will compare biomarkers on tissue, serum and wound fluid from patients with non-healing ulcers and hidradenitis to identify angiogenic and vasculogenic pathways that are dysregulated in patients with wound healing problems.

CONTACTS AND LOCATIONS:
Overall Officials: Victoria K Shanmugam, MD, Principal Investigator — George Washington University
Locations (1):
- George Washington University, Washington D.C., District of Columbia, United States